CLINICAL TRIAL: NCT01683890
Title: Incidence and Pattern of Overactive Bladder Symptoms Occurring After Hysterectomy
Brief Title: Study on Bladder and Sexual Function Change After Simple Hysterectomy
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Asan Medical Center (Other)
Collaborators: Astellas Pharma Inc (Industry)
Responsible Party: Principal Investigator, Hee-Dong Chae, Professor, Asan Medical Center
Other Study IDs: SBSFSH
Record Dates: First submitted 2012-09-04; First posted 2012-09-12 (Estimated); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Benign Uterine Disease
Keywords: Bladder symptoms; Sexual function; Quality of life; Simple hysterectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Simple hysterectomy group: Patients will undergo simple hysterectomy due to benign uterine disease.

SUMMARY:
To evaluate the incidence and pattern of bladder symptoms and sexual function change occuring after simple hysterectomy and to analyze the influence of bladder symptoms and sexual function change on quality of life of patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients who is planed to undergo simple hysterectomy due to benign uterine disease

  1. Uterine leiomyoma
  2. Uterine adenomyosis
  3. Endometrial hyperplasia
  4. Cervical intraepithelial neoplasia (including carcinoma in situ, FIGO stage IA1 cancer)
  5. Dysfunctional uterine bleeding
  6. Other benign uterine disease requiring hysterectomy

Exclusion Criteria:

* Patients who are taking medication for overactive bladder
* Patients who underwent incontinence surgery due to urinary incontinence
* Acute or chronic infectious disease of urinary tract
* Neurologic disease causing urinary abnormality
* Previous pelvic radiation therapy
* Patients who are undergoing incontinence surgery with hysterectomy
* Pregnant woman

Ages: 20 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patinets who undergo simple hysterectomy due to benign uterine disease at university hospital
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2012-09; Primary Completion 2017-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Incidence of bladder symptoms | within 6 months after surgery

SECONDARY OUTCOMES:
Pattern change of bladder symptoms after surgery | Baseline and within 6 months after surgery
Sexual function change | Baseline and within 6 months after surgery
Quality of life | within 6 months aftr surgery

CONTACTS AND LOCATIONS:
Overall Officials: Hee-Dong Chae, M.D., Ph.D., Principal Investigator — Asan Medical Center
Locations (1):
- Department of Obstetrics and Gynecology, University of Ulsan College of Medicine, Asan Medical Center, Seoul, South Korea